CLINICAL TRIAL: NCT01615835
Title: Mapping in the Coronary Sinus During Implant of a Bi-Ventricular Implantable Cardioverter Defibrillator Utilizing the NavX Mapping System
Brief Title: EnSite NavX-Guided Coronary Sinus Mapping During CRT Implant
Acronym: Bi-VNavX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 067.3
Record Dates: First submitted 2007-12-21; First posted 2012-06-11 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: EnSite NavX System — EnSite NavX system is a 3D Mapping system

SUMMARY:
Use of the EnSite NavX system to map the coronary vasculature during CRT implant

DETAILED DESCRIPTION:
Objective(s):

To determine the feasibility of CS mapping with NavX during Biventricular Implantable Cardioverter Defibrillator (BiV ICD) implantation.

Inclusion Criteria:

* Subject is between the age of 18 and 75 years
* Subject is willing and able to sign a study specific informed consent
* Subject is able to fulfill study requirements
* Meet the conventional criteria for implant of a BiV ICD, including; LVEF of ≤35%, QRS ≥ 120 ms and NYHA III-IV
* Have persistent CHF symptoms despite contemporary CHF medical therapy
* Stable and optimal medical therapy (stability is no changes in past 3 months).
* Documented history of ischemic or non-ischemic cardiomyopathy.

Exclusion Criteria:

* Have any standard device exclusions including tricuspid valve prosthesis/ replacement.
* Have a positive urine or serum pregnancy test (if female and of childbearing potential)
* Be currently participating in an IDE or IND study.

ELIGIBILITY:
Inclusion Criteria:

* Meet criteria for CRT implant including EF<35%, QRS>120ms, NYHA class III or IV
* Persistent CHF symptoms despite optimization
* Stable/optimal medical therapy
* History of ischemic or non-ischemic cardiomyopathy

Exclusion Criteria:

* Any standard device exclusion including TVR
* Positive pregnancy test
* Currently participating in IDE/IND study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-04; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Determine feasibility of CS mapping with EnSite NavX during CRT implant | Procedural

CONTACTS AND LOCATIONS:
Overall Officials: Adam Berman, MD, Principal Investigator — Augusta University
Locations (2):
- United States (2):
  - Medical College of Georgia, Augusta, Georgia
  - Duke Medical Center, Durham, North Carolina